CLINICAL TRIAL: NCT03139864
Title: Comparison of the Use of Energy Substrates and Hormonal Regulation of Blood Sugar During Exercise of Increasing Intensity Between Children With Type 1 Diabetes and Non-diabetic Control Children.
Acronym: DIABSPORT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0292; 2016-A01837-44 (Other: 2016-A01837-44)
Record Dates: First submitted 2017-04-07; First posted 2017-05-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Control; Physical activity; Substrate utilization; Hormonal regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Masking Description: no masking is used. All involved know the identity of the intervention assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- type 1 diabetes (Experimental): Comparison between infants with type 1 diabetes and infants without type 1 diabetes during exercise :
  Interventions: Procedure: controlled physical activity
- without type 1 diabetes (Active Comparator): Comparison between infants with type 1 diabetes and infants without type 1 diabetes during exercise :
  Interventions: Procedure: controlled physical activity

INTERVENTIONS:
Procedure: controlled physical activity — Comparison between infants with type 1 diabetes and infants without type 1 diabetes during exercise :

SUMMARY:
The type 1 diabetes is a common chronic disease characterised by the stop of production of insulin by the pancreas. A lot of factors modify blood glucose. The objective is to study the effect of type 1 diabetes on the use of energy substrates (fats and carbohydrates) during exercise of increasing intensity by a comparison with non-diabetic controls children.

DETAILED DESCRIPTION:
The type 1 diabetes is a common chronic disease characterised by the stop of production of insulin by the pancreas. A lot of factors modify blood glucose. The objective is to study the effect of type 1 diabetes on the use of energy substrates (fats and carbohydrates) during exercise of increasing intensity by a comparison with non-diabetic controls children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 12 years
* Tanner stage <T2
* Type 1 diabetes for more than 1 year for infants with type 1 diabetes

Exclusion Criteria:

* Tanner stage > ou = T2
* Obesity
* Hormonal disease
* Disease who prevent doing exercise

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of substrate utilization between infants with type 1 diabetes and infants without type 1 diabetes during exercise | at day 1
  Measurements will be carried out by indirect calorimetry and the relationship between CO2 et O2 (Metamax)

SECONDARY OUTCOMES:
hormonal regulation of blood glucose | at day 1
  insulin, glucagon, adrenaline, cortisol and growth hormone will be metered according to their half life until 2 hours after physical activity (T12, T20, T40, T60, T120)
lipoxmax : the intensity for wich lipid oxydation is maximum will be carried out by indirect calorimetry | at day 1
  during exercise
Comparison between infants during 10 days before and 4 days after exercise of blood glucose modification | 10 days before and 4 days after exercise of blood glucose modification
  Comparison of curves of interstitial blood glucose measured with Freestyle®

CONTACTS AND LOCATIONS:
Overall Officials: Daniel TERRAL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France